CLINICAL TRIAL: NCT01749020
Title: Effect of Polyphenol-rich Dark Chocolate on Insulin Sensitivity in Normal Weight and Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Margaret University (Other)
Collaborators: Barry Callebaut (Unknown)
Responsible Party: Principal Investigator, Grace Farhat, PhD research student, Queen Margaret University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DC-Ins01
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Insulin Resistance
Keywords: Diabetes type II, Insulin sensitivity
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyphenol-rich Dark chocolate (Experimental): Dark chocolate with 500 mg of polyphenols
  Interventions: Other: Polyphenol-rich Dark chocolate
- Placebo Dark chocolate (Placebo Comparator): This chocolate contains little or no polyphenols
  Interventions: Other: Placebo Dark chocolate

INTERVENTIONS:
Other: Polyphenol-rich Dark chocolate — Participants will be asked to consume 20g of dark chocolate containing 500mg of polyphenols daily for a period of 4 weeks
  Arms: Polyphenol-rich Dark chocolate
Other: Placebo Dark chocolate — Participants will be asked to consume 20g of dark chocolate containing little or no polyphenols for a period of 4 weeks
  Arms: Placebo Dark chocolate

SUMMARY:
The purpose of the study is to determine the effect of polyphenol-rich dark chocolate on insulin sensitivity in normal weight and overweight adults.

DETAILED DESCRIPTION:
Polyphenols may have several favourable effects on health. Dark chocolate (DC) is one of the highest sources of polyphenols in foods. The aim of the study is to determine the effect of polyphenol-rich dark chocolate on insulin sensitivity in normal weight and overweight adults. Seventy four volunteers with no history of hypertension, cardiovascular diseases or diabetes will be recruited. Participants will randomly receive 20g daily of one of the two different types of DC: Placebo DC (low in polyphenols) or DC rich in polyphenols (500mg) for a period of four weeks. Participants will be asked to make two appointments to the university clinical lab. Anthropometric measurements (height, weight, waist circumference), blood and saliva samples will be taken during each of the 2 visits. Compliance will be tested by the measure of total polyphenols in a 24-hour urine sample in some random samples before and at the end of the intervention. To monitor any fluctuations in the participants' diet or physical activity during the study period, a three-day diet diary and a physical activity questionnaire will be collected before the start of the study and after four weeks. Data will be analysed with an ANCOVA with time (pre- and post-) and treatment (DC and placebo) as between-subject factor.

ELIGIBILITY:
Inclusion Criteria:

* Adults with no history of hypertension, diabetes and cardiovascular diseases
* BMI from 18-24.9 and BMI >25
* Males and Females
* Age: 18-65 years

Exclusion Criteria:

* Participants with cardiovascular diseases, hypertension or diabetes
* Smokers and heavy alcohol drinkers
* Participants taking any medications that affect insulin, cholesterol, triglycerides or blood pressure
* Participants taking dietary supplements containing high doses of antioxidants
* Postmenopausal women taking HRT (Hormone Replacement Therapy)
* Participants who recently participated or are currently on a weight management program
* Participants with regular consumption of cocoa or DC (> 1 serving/week)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Determine if the consumption of DC rich in polyphenols can induce a change in insulin sensitivity | Baseline and week 4
  Insulin sensitivity will be determined by determined by HOMA-IR (Homeostasis Model of Assessment - Insulin Resistance)

SECONDARY OUTCOMES:
Determine if the consumption of DC rich in polyphenols can induce a change in glucose levels | Baseline and week 4
Determine if the consumption of DC rich in polyphenols can induce a change in Lipid profile (TC, HDL, LDL & TG) | Baseline and week 4
Determine if the consumption of DC rich in polyphenols can induce a change in oxidized LDL levels | Baseline and week 4
Determine if the consumption of DC rich in polyphenols can induce a change in BMI and Waist circumference | Baseline and week 4
Determine if the consumption of DC rich in polyphenols can induce a change in blood pressure | Baseline and week 4
Determine if the consumption of DC rich in polyphenols can induce a change in salivary cortisol-to-cortisone ratio | Baseline and week 4
Determine if the consumption of DC rich in polyphenols can induce a change in high sensitivity CRP | Baseline and Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Emad Al-Dujaili, PhD, Study Director — Queen Margaret University
Locations (1):
- Queen Margaret University Lab, Musselburgh, East Lothian, United Kingdom